CLINICAL TRIAL: NCT00028886
Title: A Randomized Phase III Study On The Effect Of Thalidomide Combined With Adriamycin, Dexamethasone (AD) And High Dose Melphalan In Patients With Multiple Myeloma
Brief Title: Combination Chemotherapy With or Without Thalidomide in Treating Patients With Multiple Myeloma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Commissie Voor Klinisch Toegepast Onderzoek (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000069144; CKTO-2001-02; HOVON-50MM; EU-20133; HOVON-CKVO-2001-02
Record Dates: First submitted 2002-01-04; First posted 2003-01-27 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2012-10

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Filgrastim; Interferon-alpha; Cyclophosphamide; Dexamethasone; Doxorubicin; Melphalan; Thalidomide; Vincristine; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: filgrastim
Biological: recombinant interferon alfa
Drug: cyclophosphamide
Drug: dexamethasone
Drug: doxorubicin hydrochloride
Drug: melphalan
Drug: thalidomide
Drug: vincristine sulfate
Procedure: bone marrow ablation with stem cell support
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Thalidomide may stop the growth of cancer cells by stopping blood flow to the cancer. Peripheral blood stem cell transplant using stem cells from the patient or a donor may be able to replace immune cells that were destroyed by chemotherapy used to kill cancer cells. The donated stem cells may also help destroy any remaining cancer cells (graft-versus-tumor effect). It is not yet known whether chemotherapy followed by peripheral blood stem cell transplant is more effective with or without thalidomide in treating multiple myeloma.

PURPOSE: This randomized phase III trial is studying giving combination chemotherapy with thalidomide to see how well it works compared with giving combination chemotherapy without thalidomide in treating patients with multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of doxorubicin, dexamethasone, and high-dose melphalan with versus without thalidomide, in terms of event-free survival, of patients with multiple myeloma.
* Determine the response rate, complete response rate, overall survival, and progression-free survival of patients treated with these regimens.
* Determine the safety and toxicity of thalidomide in combination with intensive chemotherapy in these patients.
* Assess the value of prognostic factors at diagnosis in individual patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center and treatment policy (1 course vs 2 courses of high-dose melphalan). Patients are randomized to 1 of 2 treatment arms.

Arm I:

* Patients receive induction chemotherapy (AD) comprising doxorubicin IV on days 1-4 and oral dexamethasone on days 1-4, 9-12, and 17-20. Patients receive oral thalidomide daily beginning on day 1 and continuing until 2 weeks before start of stem cell mobilization. Treatment repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity.
* Patients receive stem cell mobilization with chemotherapy comprising cyclophosphamide IV on day 1 and doxorubicin IV and oral dexamethasone on days 1-4 (CAD). Patients also receive filgrastim (G-CSF) subcutaneously (SC) beginning on day 5 and continuing until last apheresis.
* Beginning 8-10 weeks after stem cell collection, patients receive low-dose oral thalidomide daily and high-dose melphalan IV on days -3 and -2 as intensification. Patients undergo stem cell infusion on day 0. Patients may receive a second course of high-dose melphalan 2-3 months after the first course, in which case, stem cell infusion follows the second course of melphalan.
* Patients receive maintenance therapy with oral thalidomide daily until disease progression or after 3 months if no response.
* Beginning 2 months after the last course, patients with an HLA-identical sibling donor undergo nonmyeloablative stem cell transplantation after radiotherapy.

Arm II:

* Patients receive induction chemotherapy (VAD) comprising vincristine IV and doxorubicin IV on days 1-4 and dexamethasone on days 1-4, 9-12, and 17-20. Treatment repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity.
* Patients receive stem cell mobilization with CAD chemotherapy as in arm I. G-CSF is given as in arm I.
* Patients receive high-dose melphalan and undergo stem cell infusion as in arm I.
* Patients receive maintenance therapy with interferon alfa SC 3 times weekly until progression or after 3 months if no partial response.
* Beginning 2 months after the last course, patients with an HLA-identical sibling donor undergo nonmyeloablative stem cell transplantation after radiotherapy.

All patients are followed every 6 months for 3 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 450 patients (225 per treatment arm) will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed multiple myeloma

  * Stage II or III
* No systemic amyloid light-chain amyloidosis

PATIENT CHARACTERISTICS:

Age:

* 18 to 65

Performance status:

* WHO 0-3

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* No significant hepatic dysfunction*
* Bilirubin less than 1.75 mg/dL*
* AST/ALT less than 2.5 times normal* NOTE: *Unless related to myeloma

Renal:

* Not specified

Cardiovascular:

* No severe cardiac dysfunction
* No New York Heart Association class II, III, or IV heart disease

Other:

* HIV negative
* No active uncontrolled infection
* No other malignancy within the past 5 years except basal cell skin cancer or carcinoma in situ of the cervix
* No known intolerance to thalidomide
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Patients 18 to 55 years of age must not have been allocated before study randomization to allogeneic stem cell transplantation with an HLA-identical sibling donor

Chemotherapy:

* No more than 2 prior courses of melphalan and prednisone therapy for local myeloma progression
* No other prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* Prior local radiotherapy for local myeloma progression allowed
* No other prior radiotherapy

Surgery:

* Not specified

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2001-03

PRIMARY OUTCOMES:
Event-free survival

SECONDARY OUTCOMES:
Partial response and complete response
Overall survival
Progression-free survival
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: H. Lokhorst, MD, PhD, Study Chair — UMC Utrecht
Locations (17):
- U.Z. Gasthuisberg, Leuven, Belgium
- Netherlands (16):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Meander Medisch Centrum, Amersfoort
  - Netherlands Cancer Institute - Antoni van Leeuwenhoek Hospital, Amsterdam
  - Vrije Universiteit Medisch Centrum, Amsterdam
  - Academisch Medisch Centrum at University of Amsterdam, Amsterdam
  - Medisch Spectrum Twente, Enschede
  - University Medical Center Groningen, Groningen
  - Medisch Centrum Leeuwarden - Zuid, Leeuwarden
  - Leiden University Medical Center, Leiden
  - Academisch Ziekenhuis Maastricht, Maastricht
  - Sint Antonius Ziekenhuis, Nieuwegein
  - Universitair Medisch Centrum St. Radboud - Nijmegen, Nijmegen
  - Daniel Den Hoed Cancer Center at Erasmus Medical Center, Rotterdam
  - HagaZiekenhuis - Locatie Leyenburg, The Hague
  - University Medical Center Utrecht, Utrecht
  - Isala Klinieken - locatie Sophia, Zwolle

REFERENCES:
- [Background] Johnson DC, Corthals S, Ramos C, Hoering A, Cocks K, Dickens NJ, Haessler J, Goldschmidt H, Child JA, Bell SE, Jackson G, Baris D, Rajkumar SV, Davies FE, Durie BG, Crowley J, Sonneveld P, Van Ness B, Morgan GJ. Genetic associations with thalidomide mediated venous thrombotic events in myeloma identified using targeted genotyping. Blood. 2008 Dec 15;112(13):4924-34. doi: 10.1182/blood-2008-02-140434. Epub 2008 Sep 19. PMID 18805967
- [Result] Lokhorst HM, van der Holt B, Cornelissen JJ, Kersten MJ, van Oers M, Raymakers R, Minnema MC, Zweegman S, Janssen JJ, Zijlmans M, Bos G, Schaap N, Wittebol S, de Weerdt O, Ammerlaan R, Sonneveld P. Donor versus no-donor comparison of newly diagnosed myeloma patients included in the HOVON-50 multiple myeloma study. Blood. 2012 Jun 28;119(26):6219-25; quiz 6399. doi: 10.1182/blood-2011-11-393801. Epub 2012 Mar 22. PMID 22442350
- [Result] Lokhorst HM, van der Holt B, Zweegman S, Vellenga E, Croockewit S, van Oers MH, von dem Borne P, Wijermans P, Schaafsma R, de Weerdt O, Wittebol S, Delforge M, Berenschot H, Bos GM, Jie KS, Sinnige H, van Marwijk-Kooy M, Joosten P, Minnema MC, van Ammerlaan R, Sonneveld P; Dutch-Belgian Hemato-Oncology Group (HOVON). A randomized phase 3 study on the effect of thalidomide combined with adriamycin, dexamethasone, and high-dose melphalan, followed by thalidomide maintenance in patients with multiple myeloma. Blood. 2010 Feb 11;115(6):1113-20. doi: 10.1182/blood-2009-05-222539. Epub 2009 Oct 30. PMID 19880501
- [Result] Lokhorst HM, Schmidt-Wolf I, Sonneveld P, van der Holt B, Martin H, Barge R, Bertsch U, Schlenzka J, Bos GM, Croockewit S, Zweegman S, Breitkreutz I, Joosten P, Scheid C, van Marwijk-Kooy M, Salwender HJ, van Oers MH, Schaafsma R, Naumann R, Sinnige H, Blau I, Delforge M, de Weerdt O, Wijermans P, Wittebol S, Duersen U, Vellenga E, Goldschmidt H; Dutch-Belgian HOVON; German GMMG. Thalidomide in induction treatment increases the very good partial response rate before and after high-dose therapy in previously untreated multiple myeloma. Haematologica. 2008 Jan;93(1):124-7. doi: 10.3324/haematol.11644. PMID 18166796